CLINICAL TRIAL: NCT00381589
Title: Treatment of Clozapine-Induced Hypersalivation Ipratropium Bromide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Dr. Gary Remington, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 150/2006
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Hypersalivation
Keywords: clozapine-induced hypersalivation
MeSH Terms: conditions — Sialorrhea | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Random assignment to investigational spray
  Interventions: Drug: ipratropium bromide 0.03% spray

INTERVENTIONS:
Drug: ipratropium bromide 0.03% spray

SUMMARY:
Hypersalivation (Too much saliva) and drooling is a side effect experienced by 31% of people taking the antipsychotic clozapine. This study aims to determine if using the medication ipratropium bromide(IPB)at bedtime will reduce the amount of salivation and the distress people may feel.

DETAILED DESCRIPTION:
With the recent questions regarding the effectiveness of newer atypical antipsychotic medications in treating schizophrenia, clozapine continues to remain the gold standard for treatment-refractory schizophrenia. However, treatment with clozapine continues to be limited by its many side effects. The second most common side effect, occurring in 31% of clozapine treated patients, is hypersalivation or sialorrhea. Sialorrhea can be profoundly stigmatizing and functionally disabling in certain patients, and may increase discontinuation rates in this high-risk patient population. Several studies have evaluated the efficacy of anticholinergic agents mainly in small, uncontrolled studies or anecdotal reports and are often complicated by difficulties in medication administration and systemic side effects. Open label and case series studies have demonstrated promising results with ipratropium bromide (IPB) treatment of clozapine-induced hypersalivation, acting on anticholinergic receptors with minimal systemic absorption. However, no randomized controlled trials have evaluated IPB in the treatment of this problematic side effect.The primary goals of this study is to determine the efficacy of ipratropium bromide in reducing clozapine-induced hypersalivation, as per the Toronto Nocturnal Hypersalivation Scale, which is a modified hypersalivation scale incorporating the Drooling Severity Scale and the Nocturnal Hypersalivation Rating Scale, and reduced measurements on visual analogue scales for hypersalivation distress and severity. Our hypothesis that Ipratropium bromide use at bedtime will result in a significant reduction in nocturnal clozapine-induced hypersalivation as measured by the Toronto Nocturnal Hypersalivation Scale (TNHS) through its local anticholinergic activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder as per DSM IV-TR criteria
* Receiving clozapine for at least 2 months
* No change in their clozapine dose for at least 2 weeks
* Have a Clinical Global Impression scale score for hypersalivation of greater than or equal to 4
* Have the capacity to provide voluntary, informed consent
* Able to speak English
* Have a minimum score of 2 on the TNHS prior to study entry
* No change in medications for at least 2 weeks

Exclusion Criteria:

* Subjects with co-morbid medical conditions that could influence hypersalivation (e.g. Idiopathic Parkinson's Disease)
* Subjects currently receiving ipratropium bromide for the treatment of hypersalivation or other medical conditions
* History of narrow-angle glaucoma, prostatic hyperplasia or bladder neck obstruction
* History of an allergic reaction to ipratropium bromide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Toronto Nocturnal Hypersalivation Scale scores | intermittent
Visual Analogue Scale - Severity | intermittent
Visual Analogue Scale - Distress | Intermittent
Simpson-Angus Rating Scale | Each study visit
Clinical Global Improvement Scale | Each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sockalingam S, Shammi C, Remington G. Treatment of clozapine-induced hypersalivation with ipratropium bromide: a randomized, double-blind, placebo-controlled crossover study. J Clin Psychiatry. 2009 Aug;70(8):1114-9. doi: 10.4088/JCP.08m04495. PMID 19758522
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research